CLINICAL TRIAL: NCT03969108
Title: Diagnostic Accuracy Study of Indocyanine Green for Parathyroid Perfusion Assessment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-5447
Record Dates: First submitted 2019-05-24; First posted 2019-05-31 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Thyroid Cancer; Thyroid Goiter; Graves Disease
Keywords: Thyroid surgery; Indocyanine green (ICG); Hypoparathyroidism
MeSH Terms: conditions — Thyroid Neoplasms; Goiter; Graves Disease; Hypoparathyroidism | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Indocyanine Green (Experimental)
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — ICG is a fluorescent dye which binds tightly to plasma proteins and becomes confined to the vascular system.

SUMMARY:
This study aims to develop a standardized universal imaging protocol for ICG-guided fluorescent total thyroidectomy, including quantitative evaluations of the fluorescent signal. Therefore, patients will undergo thyroid surgery (total thyroidectomy) with the use of ICG fluorescence.

DETAILED DESCRIPTION:
Background Thyroid surgery volume continues to increase worldwide over the past few decades. During a total thyroidectomy (TTx), the ultimate goal is to remove all thyroid tissue, whereas damage to adjacent tissue is prevented. However, iatrogenic hypoparathyroidism, as a result of surgical removal or damage to the parathyroid glands, occurs in approximately 30% of the cases. In 2016 near-infrared fluorescence guided surgery with indocyanine green (ICG) was proposed for visualizing viability and blood supply of parathyroid glands during TTx. ICG can visualize tissue perfusion, since it becomes completely and permanently fixed to plasma proteins once in the bloodstream, and circulates in the intravascular compartment only. However, one of the limitations of ICG imaging is the subjectivity of the interpretation of fluorescence, which makes the assessment of images inconsistent among studies. There is a clear need for standardization of the evaluation of the perfusion with ICG, since visual evaluation of the fluorescent signal of ICG is not sufficient to reliably predict the perfusion of parathyroid glands.

Main research question To develop a standardized universal imaging protocol for ICG-guided fluorescent total thyroidectomy including quantitative evaluations of the fluorescent signal.

Design This will be a proof-of-concept , prospective cohort study of patients undergoing a total thyroidectomy with ICG-guided fluorescent surgery to evaluate tissue perfusion The main study endpoint is quantification of the fluorescent signal of ICG. Secondary outcomes are data from surgery, postoperative lab values (including calcium, PTH, albumin) and postoperative medication use.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years
2. Patients undergoing total thyroidectomy as surgical procedure for thyroid cancer, Graves' disease or goiter
3. Patients are eligible for surgery
4. Patients are mentally competent and are able and willing to comply with study procedures
5. Written informed consent

Exclusion Criteria:

1. Patients with a known allergy to ICG or iodinated contrast
2. Pregnant or lactating women
3. Patients with previous neck surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Quantification of the fluorescent signal of ICG | At time of surgery
  Quantification of the fluorescent signal of ICG

SECONDARY OUTCOMES:
Appearance of parathyroid gland | At time of surgery
  Vascularization appearance of parathyroid gland intraoperatively (1= surgeon thinks parathyroid gland is well vascularized, 2 = surgeons thinks parathyroid gland is devascularized)
Duration of surgery | From start to end of surgery
  Duration of surgery in minutes
Postoperative calcium concentration | Postoperative day 1 and at the first out-patient clinic visit (between 2 to 30 days postoperative)
  Postoperative albumin-corrected calcium concentration in blood
Postoperative PTH concentration | Postoperative day 1 and at the first out-patient clinic visit (between 2 to 30 days postoperative)
  Postoperative PTH concentration in blood
Rate of prescribed postoperative calcium medication | Postoperative day 1 and at the first out-patient clinic visit (between 2 to 30 days postoperative)
  Rate of prescribed postoperative calcium medication
Rate of prescribed postoperative vitamin D medication | Postoperative day 1 and at the first out-patient clinic visit (between 2 to 30 days postoperative)
  Rate of prescribed postoperative vitamin D medication

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Pasternak, MD, MPHc, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No